CLINICAL TRIAL: NCT02014909
Title: Part I and Part II A Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of KTN3379 in Adult Subjects With Advanced Tumors Alone or With Chemotherapy
Brief Title: A Phase 1 Study to Evaluate the Safety and Pharmacokinetics of KTN3379 in Adult Subjects With Advanced Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTN3379-CL-001
Record Dates: First submitted 2013-12-04; First posted 2013-12-18 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Advanced Cancer
Keywords: KTN3379; Advanced cancer; Phase 1; Monoclonal antibody; Safety and pharmacokinetics; CDX3379

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- KTN3379 (Experimental): KTN3379
  Interventions: Biological: KTN3379
- Part II, Arm A (Experimental): Combination of KTN3379 and cetuximab
  Interventions: Biological: KTN3379
- Part II, Arm B (Experimental): Combination of KTN3379 and erlotinib
  Interventions: Biological: KTN3379
- Part II, Arm C (Experimental): Combination of KTN3379 and vemurafenib
  Interventions: Biological: KTN3379
- Part II, Arm D (Experimental): Combination of KTN3379 and trastuzumab
  Interventions: Biological: KTN3379

INTERVENTIONS:
Biological: KTN3379 — Single agent KTN3379 or in combination administered until unacceptable toxicity or progressive disease

SUMMARY:
Part I will evaluate the pharmacokinetic profile and safety of KTN3379 over several doses with the objective of defining a Phase 2 dose in patients with advanced malignancies. Part II will evaluate the pharmacokinetic profile and safety of KTN3379 in combination with other targeted agents and obtain preliminary evidence of anti tumor activity in specific types of cancer. Patients will continue receiving KTN3379 alone or in combination until disease progression or toxicity that necessitates discontinuation (whichever comes first).

ELIGIBILITY:
Major Inclusion Criteria:

* Part I Histologically- or cytologically-confirmed advanced solid tumors that are refractory to standard therapy or for which no standard therapy exist. Part II Arm A have head and neck cancer or K-Ras wild type EGFR expressing colon cancer, Arm B, have non small cell lung cancer, Arm C, have BRAF V600E mutated melanoma and Arm D have HER2 positive breast or gastric cancer that has progressed following one or more treatments for advanced or metastatic disease.
* Eastern Cooperative Oncology Group (ECOG) status of 0 or 1
* Adequate organ function as defined below:

  * Hemoglobin ≥ 9 g/dL
  * Absolute neutrophil count ≥ 1500/mm3
  * Platelet count ≥ 100,000/mm3
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 × institutional upper limit of normal (ULN) for cases involving liver metastasis and ≤ 2.5 ×ULN for all other cases
  * Bilirubin ≤ 1.5 × ULN except for cases of documented or suspected Gilbert's disease, in which bilirubin must be ≤ 5 × ULN
  * Serum creatinine ≤ 1.5 g/dL
* Measurable disease by RECIST
* Females must be surgically sterile, one year post menopausal or negative results for a pregnancy test performed at Screening and agree to use two methods of contraception; Males who have not had a vasectomy must agree to two methods of contraception

Major Exclusion Criteria:

* Receipt of anticancer therapy:

  * within 3 weeks prior to the first dose of KTN3379, or
  * within 6 weeks or 7 half lives prior to the first dose of KTN3379 in the case of anticancer therapy involving MAbs, or
  * within 2 weeks prior to the first dose of KTN3379 in the case of palliative radiation therapy.
* Symptomatic or untreated central nervous system metastases requiring concurrent treatment, including but not limited to surgery, radiation, and/or corticosteroids; if treated, subject must be asymptomatic for 3 months prior to study entry
* Subjects who are known to have a history of or active human immunodeficiency virus (HIV) or active hepatitis B and/or C
* Uncontrolled intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, uncontrolled or idiopathic hypotension, unstable angina pectoris, cardiac arrhythmia including atrial fibrillation, active peptic ulcer disease or gastritis, or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results
* Subjects with a left ventricular cardiac ejection fraction < 50% as assessed by an echocardiogram or MUGA scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-01; Primary Completion 2017-05-25 (Actual); Study Completion 2017-06-05 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities for KTN3379 alone or in combination | Participants will be followed for the duration of treatment, an expected average of 3 cycles/9 weeks
  Continued assessment of safety

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC 0 through end of study) | Prior to the initial dose on day 1 through duration of treatment, an expected average of 3 cycles/9 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Sarah Cannon Research Institute, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee